CLINICAL TRIAL: NCT03816358
Title: A Phase I Study of Anetumab Ravtansine in Combination With Either Anti-PD-1 Antibody, or Anti-CTLA4 and Anti-PD-1 Antibodies or Anti-PD-1 Antibody and Gemcitabine in Mesothelin-Positive Advanced Pancreatic Adenocarcinoma
Brief Title: Testing the Combination of Anetumab Ravtansine With Either Nivolumab, Nivolumab and Ipilimumab, or Gemcitabine and Nivolumab in Advanced Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-00242; NCI-2019-00242 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PJC-026; 10208 (Other: University Health Network Princess Margaret Cancer Center LAO); 10208 (Other: CTEP); UM1CA186644 (NIH)
Record Dates: First submitted 2019-01-24; First posted 2019-01-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Adenocarcinoma; Stage II Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — anetumab ravtansine; Biopsy; Specimen Handling; Gemcitabine; Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (anetumab ravtansine, nivolumab) (Experimental): Patients receive anetumab ravtansine IV over 1 hour on day 1 and nivolumab IV over 30 minutes on day 8 of cycle 1 and on day 1 of subsequent cycles. Treatment repeats every 21 or 28 days (cycle 1) for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo a biopsy and collection of blood on study.
  Interventions: Biological: Anetumab Ravtansine; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Biological: Nivolumab
- Arm II (anetumab ravtansine, nivolumab, ipilimumab) (Experimental): Patients receive anetumab ravtansine IV over 1 hour on day 1 and nivolumab IV over 30 minutes on day 8 of cycle 1 and on day 1 of subsequent cycles. Patients also receive ipilimumab IV over 30 minutes on day 8 of cycle 1 and on day 1 of cycles 2-4. Treatment repeats every 21 or 28 days (cycle 1) for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo a biopsy and collection of blood on study.
  Interventions: Biological: Anetumab Ravtansine; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Biological: Ipilimumab; Biological: Nivolumab
- Arm III (anetumab ravtansine, nivolumab, gemcitabine) (Experimental): Patients receive anetumab ravtansine IV over 1 hour on day 1 and nivolumab IV over 30 minutes on day 8 of cycle 1 and on day 1 of subsequent cycles. Patients also receive gemcitabine hydrochloride over 30-40 minutes on days 1 and 8. Treatment repeats every 21 or 28 days (cycle 1) for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo a biopsy and collection of blood on study.
  Interventions: Biological: Anetumab Ravtansine; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Gemcitabine Hydrochloride; Biological: Nivolumab

INTERVENTIONS:
Biological: Anetumab Ravtansine — Given IV
  Other Names: BAY 94-9343
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
  Arms: Arm III (anetumab ravtansine, nivolumab, gemcitabine)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Arm II (anetumab ravtansine, nivolumab, ipilimumab)
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase I trial studies the side effects and best dose of anetumab ravtansine when given together with nivolumab, ipilimumab and gemcitabine hydrochloride in treating patients with mesothelin positive pancreatic cancer that has spread to other places in the body (advanced). Anetumab ravtansine is a monoclonal antibody, called anetumab ravtansine, linked to a chemotherapy drug called DM4. Anetumab attaches to mesothelin positive cancer cells in a targeted way and delivers DM4 to kill them. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving anetumab ravtansine together with nivolumab, ipilimumab, and gemcitabine hydrochloride may work better in treating patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of anetumab ravtansine with the following combinations in patients with mesothelin positive pancreatic adenocarcinoma.

SECONDARY OBJECTIVES:

I. To assess the preliminary anti-tumor activity of anetumab ravtansine (anetumab) in combination with nivolumab, nivolumab and ipilimumab, nivolumab and gemcitabine hydrochloride (gemcitabine) as measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 overall response rate (ORR).

II. To characterize the pharmacokinetics (PK) profile of anetumab (apparent diffusion coefficient [ADC]), total antibody (ADC and cleaved free antibody), DM4 and DM4-Me (S-Methyl metabolite of DM4).

III. To evaluate the tumor microenvironment and immune changes in tumor and peripheral blood over the course of treatment to identify predictors of response or resistance to treatment.

IV. To measure the progressive disease (PD) effects of this combination including molecular and immune biomarkers in tumor biopsies and peripheral blood.

EXPLORATORY OBJECTIVES:

I. To characterize mesothelin, PD-L1, CD3, CD4, CD8 expressions at baseline and after treatment in mesothelin positive pancreatic cancer patients.

II. To evaluate level of soluble mesothelin and megakaryocyte potentiation factor (MPF) over the course of treatment and to correlate these biomarkers with clinical outcome.

III. To perform whole exome sequencing (WES) +/- ribonucleic acid sequencing (RNAseq) in the tumor biopsy specimens and correlation genomic (e.g. mutational burden) and transcriptomic biomarkers with clinical outcome.

IV. To evaluate mononuclear phagocyte system (MPS) function, Fc-gamma receptors (FcgammaRs) and hormone and chemokine mediators as methods to evaluate factors affecting the PK and PD of these agents.

V. To evaluate anti-drug antibody (ADA) titres changes pre and post treatment and correlate them with PK, toxicity and responses.

OUTLINE: This is a dose-escalation study of anetumab ravtansine. Patients are assigned to 1 of 3 arms.

ARM I: Patients receive anetumab ravtansine intravenously (IV) over 1 hour on day 1 and nivolumab IV over 30 minutes on day 8 of cycle 1 and on day 1 of subsequent cycles. Treatment repeats every 21 or 28 days (cycle 1) for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo a biopsy and collection of blood on study.

ARM II: Patients receive anetumab ravtansine IV over 1 hour on day 1 and nivolumab IV over 30 minutes on day 8 of cycle 1 and on day 1 of subsequent cycles. Patients also receive ipilimumab IV over 30 minutes on day 8 of cycle 1 and on day 1 of cycles 2-4. Treatment repeats every 21 or 28 days (cycle 1) for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo a biopsy and collection of blood on study.

ARM III: Patients receive anetumab ravtansine IV over 1 hour on day 1 and nivolumab IV over 30 minutes on day 8 of cycle 1 and on day 1 of subsequent cycles. Patients also receive gemcitabine hydrochloride over 30-40 minutes on days 1 and 8. Treatment repeats every 21 or 28 days (cycle 1) for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo a biopsy and collection of blood on study.

After completion of study treatment, patients are followed up every 8 weeks for up to 100 days, then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed pancreatic adenocarcinoma that is metastatic or unresectable or recurrent
* Only subjects with positive mesothelin expression (Ventana mesothelin [MSLN]- immunohistochemistry [IHC]; Negative=H-score =< 10) are eligible. This is to be performed centrally. For dose escalation cohorts, patients with mesothelin expression in >= 5% of tumor cells are eligible. For dose expansion, patients must have moderate or strong tumor mesothelin expression defined as >= 30% of tumor cells with mesothelin expression of 2+/3 on immunohistochemical staining
* Patients must be >= 18 years of age
* Patients must have received and either progressed or been intolerant to at least 1 systemic therapy
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status score 0-1 (Karnofsky >= 80%)
* Prior anti-cancer treatments are permitted (i.e. chemotherapy, including gemcitabine and nab-paclitaxel; radiotherapy; hormonal, or immunotherapy with the exception of anti-CTLA4, anti-PD1/PD-L1, and combination of anti-CTLA4 and anti-PD1/PD-L1) providing toxicity (except for alopecia) related to prior anti-cancer therapy and/or surgery have either resolved, improved to baseline or G1
* At least one (1) measurable lesion at baseline by computed tomography (CT) or magnetic resonance imaging (MRI) as per RECIST version (v)1.1; measurable disease is a requirement in both dose escalation phase and dose expansion phase

  * Note: Measurable lesions may be in an irradiated field as long as there is documented progression and the lesion(s) can be reproducibly measured
* At least one lesion safely accessible for biopsy unless medically contraindicated; biopsies are mandatory both in dose escalation and in dose expansion; in dose escalation and in expansion the following biopsies are optional: at baseline and at progression; biopsy could be: core needle or excisional or punch biopsy. Irradiated lesions can be biopsied if tumor growth is confirmed
* Patients must have archival tumor tissue for mesothelin expression and correlative biomarker studies; subjects must consent to provide tumor blocks or slides and the availability of the tissue must be confirmed prior to subjects receiving study medication; if an archived tumor specimen is unavailable or unsuitable for correlative biomarker studies, a pre-treatment fresh tumor biopsy is required
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours of study enrollment or randomization; WOCBP must agree to appropriate methods of contraception for the duration of treatment and for 6 months after completion of treatment; males who are sexually active with a partner of childbearing potential must agree to appropriate methods of contraception for the duration of treatment. For all male patients, prior to treatment, advice should be sought for conserving sperm due to the chance of irreversible infertility as a consequence of treatment; genetic consultation is recommended if the patient wishes to have children after ending treatment; the investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control

  * Highly effective (failure rate of less than 1% per year) contraception methods include:

    * Combined (estrogen and progesterone containing: oral, intravaginal, transdermal) and progesterone-only (oral, injectable, implantable) hormonal contraception associated with inhibition of ovulation
    * Intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
    * Bilateral tubal occlusion or vasectomized partner (provided that partner is the sole sexual partner and has received medical assessment of the surgical success)
    * Sexual abstinence (reliability to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient)
  * Male patients with a female partner of childbearing potential must use a condom and ensure that an additional form of contraception is also used during

    * Note: a woman is considered WOCBP, i.e. fertile, following menarche and until becoming postmenopausal unless permanently sterile; permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy
  * A postmenopausal state is defined as no menses for 12 months without an alternative medical cause; a high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; a man is considered fertile after puberty unless permanently sterile by bilateral orchiectomy
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL

  * Patients must have not had a transfusion in the 2 weeks preceding this hemoglobin (Hb) measurement
* Total bilirubin =< institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Creatinine =< institutional ULN OR glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2
* Albumin >= 2.5 mg/dL
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients not recovered from clinically significant adverse events of their most recent therapy/intervention prior to enrollment. Concurrent enrollment in a non-interventional clinical study or the follow-up period of an interventional study is allowed.
* Untreated central nervous system (CNS) metastatic disease, leptomeningeal disease, or cord compression; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least six weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 14 days prior to trial treatment
* Evidence of uncontrolled, active infection, requiring parenteral anti-bacterial, anti-viral or anti-fungal therapy (washout: 7 days prior to cycle 1 day 1 [C1D1])
* Patients are prohibited from receiving the following therapies during the screening and treatment phase of this trial:

  * Antineoplastic systemic chemotherapy or biological therapy
  * Radiation therapy

    * Note: Radiation therapy to a symptomatic solitary lesion or to the brain may be considered on an exceptional case by case basis after consultation with Cancer Therapy Evaluation Program (CTEP); the patient must have clear measurable disease outside the radiated field; administration of palliative radiation therapy will be considered clinical progression for the purposes of determining progression free survival (PFS)
  * Live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial; examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Chalmette-Guerin (BCG), typhoid (oral) vaccine, and intranasal influenza vaccines (e.g., Flu-Mist)
* Current or prior use of systemic immunosuppressive medication (except corticosteroids at physiological doses, not exceeding 10 mg prednisone-equivalent day) within 10 days before the first dose of study medication; intranasal, inhaled, topical, or local steroid injections are allowed; steroids as premedication for hypersensitivity reactions (i.e. CT scan premedication) are allowed; systemic glucocorticoids used to modulate symptoms from an event of suspected immunologic etiology are permitted
* Any major surgery within 4 weeks of study drug administration
* Concomitant second malignancies (except adequately treated squamous cell carcinoma [SCC] or basal cell carcinoma [BCC] skin cancers or in situ bladder, breast or cervical cancers) within the last 3 years prior to study entry
* Uncontrolled or significant cardiovascular disease, including but not limited to ongoing or active symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, unstable cardiac arrhythmia
* National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5 >= grade (G)2 peripheral neuropathy (sensory or motor)
* Patients with corneal epitheliopathy and at the discretion of the ophthalmologist any other eye disorder

  * Note: Low grades of superficial punctate keratitis, within the range seen in the normal population, should not lead to the exclusion of the patient
* Active or prior documented inflammatory bowel disease (i.e. ulcerative colitis)
* Active or prior documented autoimmune disease within the past 2 years

  * Note: subjects with vitiligo, Grave's disease, psoriasis not requiring systemic treatment or hypothyroidism (i.e. following Hashimoto syndrome) stable on hormone replacement are not excluded
* Recent history or current evidence of bleeding disorder (i.e. any CTCAE G >= 2 hemorrhage/bleeding event within 28 days before the start of treatment)
* Active human immunodeficiency virus (HIV), hepatitis B or C infection; HIV-positive patients on antiretroviral therapy with undetectable viral load will not be excluded from the trial; subjects with treated hepatitis B or C with unquantifiable viral loads and no organ compromise are not excluded
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued for at least 6 months after last dose of study drugs; these potential risks may also apply to other agents used in this study; should a patient become pregnant or suspect she is pregnant while she is participating in this study, the patient should inform the treating physician immediately
* Participants who have had prior organ transplants (i.e. renal, lung, heart) due to the potential for increased rejection with immunotherapy
* Patients taking strong CYP3A4 inhibitors or strong CYP3A4 inducers within 2 weeks before the start of study treatment are excluded; consumption of grapefruit or its juice, and other fruit/juices which are strong CYP3A4 inhibitors within 2 weeks of study treatment is also not permitted; examples of strong CYP3A4 inhibitors include the following: indinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, nefazodone, and saquinavir; examples of strong CYP3A4 inducers include the following: carbamazepine, rifampin, phenytoin, St. John's wort, and phenobarbital; these lists are not exhaustive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 30-37 days post treatment
  This study will follow a 3+3 dose escalation design.

SECONDARY OUTCOMES:
Biomarker analysis | Up to 100 days post treatment
  The analysis on proposed biomarkers is hypothesis generating in nature. Descriptive statistics will be used for analysis of biomarkers. The key biomarker is CD8. CD8 after anetumab will be compared with CD8 after immunotherapy. Paired T-test will be carried out to identify changes in each biomarker between time points and mixed model will be used to study the trend in biomarkers over time when multiple measurements are available. The association between baseline biomarkers or change in biomarkers and clinical outcome progression-free survival, toxicity and overall response will also be analyzed by Cox model or logistic model where appropriate. The results may be adjusted using Pocock method for multiplicity.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Spreafico, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (45):
- United States (44):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/58/NCT03816358/ICF_000.pdf